CLINICAL TRIAL: NCT04113382
Title: A Randomized, Assessor-Blind, Parallel-Groups, Multicenter Trial Assessing the Safety and Efficacy, Including Pharmacokinetic Assessments, of CLENPIQ in Children Aged 2 Years to Less Than 9 Years
Brief Title: Study Assessing CLENPIQ as Bowel Preparation for Pediatric Colonoscopy
Acronym: PICCOLO
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 000359
Record Dates: First submitted 2019-10-01; First posted 2019-10-02 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-08

CONDITIONS: Bowel Preparation
Keywords: Colon Cleansing; Preparation for Colonoscopy
MeSH Terms: interventions — polyethylene glycol 3350

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Participants aged 2 to <4 years: CLENPIQ (Experimental): CLENPIQ administered using "split-dose" method and consists of two separate doses: the first dose (½ bottle [approximately 80 mL]) one day before colonoscopy between 5:00 PM and 9:00 PM, and the second dose (½ bottle [approximately 80 mL]) the next day, at least 5 hours prior but no more than 9 hours prior to the colonoscopy. Following each dose, participants will consume 50 mL/kg of clear liquids, up to a limit of 1,000 mL.
  Interventions: Drug: CLENPIQ
- Participants aged 2 to <4 years: MIRALAX (Active Comparator): MIRALAX 3.4 to 4.9 g/kg up to a maximum of 238 g is reconstituted with non-carbonated, clear beverage, or water and administered in increments of 4 ounce (oz) for every 30 minutes, one day before colonoscopy between 5:00 PM and 9:00 PM. Following dosing, participants will consume 50 mL/kg of clear liquids, up to a limit of 1,000 mL total weight-based maximum.
  Interventions: Drug: MIRALAX
- Participants aged 4 to <9 years: CLENPIQ (Experimental): CLENPIQ administered using "split-dose" method and consists of two separate doses: the first dose (1 bottle [approximately 160 mL]) one day before colonoscopy between 5:00 PM and 9:00 PM, and the second dose (½ bottle [approximately 80 mL]) the next day, at least 5 hours prior but no more than 9 hours prior to the colonoscopy. Following each dose, participants will consume 50 mL/kg of clear liquids, up to a limit of 1,000 mL total weight-based maximum.
  Interventions: Drug: CLENPIQ
- Participants aged 4 to <9 years: MIRALAX (Active Comparator): MIRALAX 3.4 to 4.9 g/kg up to a maximum of 238 g is reconstituted with non-carbonated, clear beverage, or water and administered in increments of 8 oz for every 30 minutes one day before colonoscopy between 5:00 PM and 9:00 PM. Following dosing, participants will consume 50 mL/kg of clear liquids, up to a limit of 1,000 mL total weight-based maximum.
  Interventions: Drug: MIRALAX

INTERVENTIONS:
Drug: CLENPIQ — CLENPIQ consists of sodium picosulfate 10.0 mg + magnesium oxide 3.5 g + citric acid, anhydrous 12.0 g.
  Supplied as a pre-mixed, ready-to-drink oral solution in two bottles, each containing 160 mL.
  Arms: Participants aged 2 to <4 years: CLENPIQ; Participants aged 4 to <9 years: CLENPIQ
Drug: MIRALAX — MIRALAX powder for oral solution, supplied in a 8.3 oz multi-dose bottle containing 238 g of laxative powder (polyethylene glycol [PEG] 3350).
  Arms: Participants aged 2 to <4 years: MIRALAX; Participants aged 4 to <9 years: MIRALAX

SUMMARY:
Bowel preparation for pediatric colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 2 years to <9 years being scheduled to undergo elective colonoscopy.
* Weight ≥10 kg (≥22 lbs).
* Participants must have had an average of three or more spontaneous bowel movements (SBM) per week for 1 month prior to the colonoscopy.
* Written informed consent (by parent(s)/ caregiver(s)/ guardian(s)) and assent (if applicable) obtained at screening.

Exclusion Criteria:

* History of significant liver, cardiovascular, or renal disease (including recent or ongoing oliguria).
* Acute surgical abdominal conditions (e.g., acute obstruction or perforation) during the screening period.
* Clinically significant abdominal pain during the screening period.
* Severe acute inflammatory bowel disease (IBD) during the screening period.
* Any prior colorectal surgery, excluding appendectomy and polyp removal.
* History of colon disease (e.g., Hirschsprung disease, volvulus, idiopathic pseudo-obstruction, or hypomotility syndrome).
* History of or ongoing intestinal ulceration, toxic megacolon or other toxic colitis.
* History of upper gastrointestinal disorder (e.g., active ulcer, pyloric stenosis or other cause of gastric retention, gastroparesis, or ileus).
* History of upper gastrointestinal surgery (e.g., gastric resection or gastric bypass), excluding cholecystectomy.
* Chronic or persistent, severe nausea or vomiting during the screening period.
* Moderate to severe dehydration during the screening period.
* Prior history of epileptic reaction, convulsions, or seizures.
* Any clinically relevant neurological events with or without association with hyponatremia during the screening period.
* Serum creatinine, estimated glomerular filtration rate (eGFR), potassium, or sodium outside normal limits during the screening period.
* Hypermagnesemia during the screening period.
* Use of the following prohibited medication: lithium (within 48 hours prior to procedure), laxatives (within 24 hours prior to procedure), drugs that in the opinion of the investigator are causing constipation in the participant (within 48 hours prior to procedure), antidiarrheal drugs (within 72 hours prior to procedure), or oral iron preparations (within 1 week prior to procedure).
* Participation in an interventional investigational trial requiring administration of an investigational drug within 30 days prior to receiving trial medication (or within 60 days for investigational drugs with an elimination half-life >15 days).
* Any clinically relevant abnormal findings in medical history, physical examination, vital signs, electrocardiogram (ECG), clinical chemistry, hematology, coagulation, or urinalysis at screening which in the opinion of the investigator(s), might put the participant at risk because of his/her participation in the trial.
* Hypersensitivity to any of the ingredients of the trial medications.
* Inability to comply with the dietary restrictions in the trial or the fluid requirements before and after investigational medicinal product (IMP) administration.

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants classified as responders, defined by "excellent" or "good" in the Modified Aronchick scale | On the day of colonoscopy (Day 1)
  The efficacy of overall colon cleansing in terms of responders will be graded by a blinded endoscopist using the Modified Aronchick Scale. It is a 4-point scale that grades colon cleansing as Excellent (>90% of mucosa seen, mostly liquid stool, minimal suctioning needed for adequate visualization), Good (>90% of mucosa seen, mostly liquid stool, significant suctioning needed for adequate visualization), Fair (>90% of mucosa seen, mixture of liquid and semisolid stool, could be suctioned and/or washed) or Inadequate (<90% of mucosa seen, mixture of semisolid and solid stool which could not be suctioned or washed).The participant is considered to be a responder if overall colon cleansing is "excellent" or "good" on this 4-point scale.

SECONDARY OUTCOMES:
Percentage of participants classified as "excellent" in the Modified Aronchick scale | On the day of colonoscopy (Day 1)
  The efficacy of overall colon cleansing in terms of responders will be graded by a blinded endoscopist using the Modified Aronchick Scale. It is a 4-point scale that grades colon cleansing as Excellent (>90% of mucosa seen, mostly liquid stool, minimal suctioning needed for adequate visualization), Good (>90% of mucosa seen, mostly liquid stool, significant suctioning needed for adequate visualization), Fair (>90% of mucosa seen, mixture of liquid and semisolid stool, could be suctioned and/or washed) or Inadequate (<90% of mucosa seen, mixture of semisolid and solid stool which could not be suctioned or washed). Percentage of participants classified as "excellent" in the Modified Aronchick scale will be reported.
Percentage of participants who completed the assigned dose of CLENPIQ among participants in whom nasogastric tube was not utilized to assist with CLENPIQ dosing | From randomization (Day -1) up to second dose of CLENPIQ (Day 1)
  A nasogastric tube may be inserted if the participant is likely to fail to drink the prescribed amount of cleanout preparation within the required time. Percentage of participants who completed the assigned dose of CLENPIQ without utilizing nasogastric tube will be reported.
Frequency of each category of the Modified Tolerability and Satisfaction Questionnaire: How easy was it for you/the child to drink the bowel cleanout medicine? | On the day of colonoscopy (Day 1)
  The tolerability and satisfaction of colon cleansing preparation for colonoscopy will be assessed by the child/ parent(s)/caregiver(s)/guardian(s) using modified tolerability and satisfaction questionnaire. The above question will be answered on a 6-point scale: (1=very easy, 2=easy, 3=okay, 4=difficult, 5=very difficult, 6=do not know).
Frequency of each category of the Modified Tolerability and Satisfaction Questionnaire: How did the bowel cleanout medicine taste? | On the day of colonoscopy (Day 1)
  The tolerability and satisfaction of colon cleansing preparation for colonoscopy will be assessed by the child/ parent(s)/caregiver(s)/guardian(s) using modified tolerability and satisfaction questionnaire. The above question will be answered on a 6-point scale: (1=very well, 2=well, 3=okay, 4=bad, 5=very bad, 6=do not know).
Frequency of each category of the Modified Tolerability and Satisfaction Questionnaire: How often did your/the child's tummy hurt since you/the child started the cleanout? | On the day of colonoscopy (Day 1)
  The tolerability and satisfaction of colon cleansing preparation for colonoscopy will be assessed by the child/parent(s)/caregiver(s)/guardian(s) using modified tolerability and satisfaction questionnaire. The above question will be answered on a 6-point scale: (1=never, 2=rarely, 3=sometimes, 4=often, 5=very often, 6=do not know).
Frequency of each category of the Modified Tolerability and Satisfaction Questionnaire: How often did you/the child feel fullness in your/the child's tummy since you/the child started the cleanout? | On the day of colonoscopy (Day 1)
  The tolerability and satisfaction of colon cleansing preparation for colonoscopy will be assessed by the child/ parent(s)/caregiver(s)/guardian(s) using modified tolerability and satisfaction questionnaire. The above question will be answered on a 6-point scale: (1=never, 2=rarely, 3=sometimes, 4=often, 5=very often, 6=do not know).
Frequency of each category of the Modified Tolerability and Satisfaction Questionnaire: How often did you/the child wake up last night? | On the day of colonoscopy (Day 1)
  The tolerability and satisfaction of colon cleansing preparation for colonoscopy will be assessed by the child/ parent(s)/caregiver(s)/guardian(s) using modified tolerability and satisfaction questionnaire. The above question will be answered on a 6-point scale: (1=never, 2=rarely, 3=sometimes, 4=often, 5=very often, 6=do not know).
Frequency of each category of the Modified Tolerability and Satisfaction Questionnaire: How often did you/the child feel sick to your/the child's stomach (nausea) since you/the child started the cleanout? | On the day of colonoscopy (Day 1)
  The tolerability and satisfaction of colon cleansing preparation for colonoscopy will be assessed by the child/ parent(s)/caregiver(s)/guardian(s) using modified tolerability and satisfaction questionnaire. The above question will be answered on a 6-point scale: (1=never, 2=rarely, 3=sometimes, 4=often, 5=very often, 6=do not know).
Frequency of each category of the Modified Tolerability and Satisfaction Questionnaire: How much were you/the child bothered by going to the bathroom since you/the child started the cleanout? | On the day of colonoscopy (Day 1)
  The tolerability and satisfaction of colon cleansing preparation for colonoscopy will be assessed by the child/parent(s)/caregiver(s)/guardian(s) using modified tolerability and satisfaction questionnaire. The above question will be answered on a 6-point scale: (1=never, 2=rarely, 3=sometimes, 4=often, 5=very often, 6=do not know).
Systemic concentrations of picosulfate and bis-(p-hydroxyphenyl)-pyridyl-2-methane (BHPM, active metabolite of picosulfate) after randomization | For PK1 subset: 3 to 6 hours after the second dose of CLENPIQ prior to colonoscopy (Day 1); For PK3 subset: 15 minutes before, 1 to 2 hours, and 3 to 6 hours after second dose of CLENPIQ prior to colonoscopy (Day 1)
  For the assessment of picosulfate and BHPM concentrations, participants randomized to CLENPIQ will be further randomized (1:1 ratio) for collection of either 1 pharmacokinetic (PK) sample (PK1 subset) or 3 PK samples (PK3 subset).
Systemic concentrations of magnesium at screening | Screening (≤21 days before scheduled colonoscopy)
  At screening, PK assessments of magnesium concentrations will be performed for all participants.
Systemic concentrations of magnesium after randomization | 3 to 6 hours after second dose of CLENPIQ prior to colonoscopy (Day 1); 1 or 2 days after the colonoscopy (Day 2 or 3)
  After randomisation, PK assessments of magnesium concentrations will be performed only for the participants randomized to CLENPIQ.
Percentage of participants with adverse events (AEs) | From screening (≤21 days before scheduled colonoscopy) up to Day 28±7 after colonoscopy
  An AE is defined as any untoward medical occurrence in a participant participating in a clinical study.
  Percentage of participants with any AE (serious or non-serious) will be presented.
Percentage of participants with abnormal findings in vital signs | From screening (≤21 days before scheduled colonoscopy) up to Day 28±7 after colonoscopy
  Percentage of participants with abnormal findings (clinically significant) in vital signs will be reported.
Percentage of participants with abnormal findings in clinical laboratory tests | From screening (≤21 days before scheduled colonoscopy) up to Day 28±7 after colonoscopy
  Percentage of participants with abnormal findings (clinically significant) in clinical laboratory tests will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (4):
- United States (4):
  - Ferring Investigational Site, Mobile, Alabama
  - Ferring Investigational Site, San Diego, California
  - Ferring Investigational Site, Baltimore, Maryland
  - Ferring Investigational Site, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No